CLINICAL TRIAL: NCT05929365
Title: Development and Clinical Utility of a New Method to Identify Patients With Risk of Recurrent Colorectal Lesions and Personalization of Their Surveillance Based on Mutation Burden and Clinical-pathological Phenotype
Brief Title: Innovative Approach to Detect Recurrent Colorectal Lesions With Surveillance Via Mutation Analysis & Clinical Phenotype
Acronym: MTG
Status: Recruiting | Type: Observational
Sponsor: Military University Hospital, Prague (Other)
Responsible Party: Principal Investigator, Stepan Suchanek, MD., Ph.D., Principal Investigator, Military University Hospital, Prague
Other Study IDs: NU22-08-00424
Record Dates: First submitted 2023-06-25; First posted 2023-07-03 (Actual); Last update posted 2023-07-03 (Actual); Status verified 2023-06

CONDITIONS: Predictive Cancer Model
Keywords: phenotype; surveillance; colonoscopy; colorectal neoplasia; genetic mutation; metachronous lesions
MeSH Terms: interventions — Colonoscopy; Endoscopic Mucosal Resection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Biospecimen Retention: Samples With DNA — colorectal lesions (polyps)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: colonoscopy — determine the mutation profile of resected colorectal neoplasia
  Other Names: endoscopic resection

SUMMARY:
It is known that the development of colorectal adenoma is dependent on the appearance of somatic mutations in protooncogenes and tumor suppressor genes. Based on our previous mutation analyses of 120 patients with high-risk adenoma removed by enbloc resection with subsequent colonoscopy after 1 year, there is a correlation between mutation in exon 7 of the TP53 gene and risk of early metachronous lesions development. The results also indicate that mutation phenotype (mutation profile and burden) of all lesions detected on index colonoscopy can determine risk of metachronous lesions. As not all synchronous lesions were analyzed and the surveillance colonoscopy interval was less than 3 years, this assumption could not be confirmed. In this study it is planned to perform mutation analysis of all synchronous lesions in 200 patients and correlate the data with appearance of metachronous lesions after 1, 3 and 5 years. Moreover, the mutation profile of all metachronous lesions developed during the 5 years of surveillance will be determinated and compared with mutation profile of index lesions from the same localization to verify their common biological origin. This all could help personalize the surveillance program in terms of reduction of the burden on the patient and endoscopic workplaces and risk of developing colorectal cancer in a particular patient.

DETAILED DESCRIPTION:
The aim of this prospective study is to identify patients with recurrent colorectal lesions risk and try to design an optimal intervals of surveillance colonoscopies, especially in the high-risk group of patients, using mutation and clinical-pathologic phenotype. The partial goals are: 1. Determination of the mutation profile and mutation burden in 200 patients based on examination of all their index and synchronous lesions found during index colonoscopy using an established PCR/DCE-based heteroduplex method. 2. Clinical and histopathological evaluation and mutational profiling of all metachronous lesions found during five-year surveillance period. 3. Correlation of clinical and histopathological parameters with mutational phenotype of patient. 4. Correlation of patient's mutational phenotype with an occurrence of metachronous lesion/s during surveillance period. 5. Comparison of the mutation profile of lesions from the index period withthe mutation profile of metachronous lesions. 6. Analysis of the similarity of the mutation profile of lesions found in the same / close areas of the colorectum.

ELIGIBILITY:
Inclusion Criteria:

* Colorectal polyp larger than 10mm removed by colonoscopy therapeutic method (EPE, EMR, ESD)
* Signed informed consent with the study and with colonoscopy

Exclusion Criteria:

* FAP, HNPCC and other hereditary CRC syndromes probands
* Colonoscopy contraindication
* Severe acute inflammatory bowel disease
* Severe comorbidities; likely non-compliance of the patient

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with colorectal neoplasia detected in diagnostic colonoscopy.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2022-05-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Development and Clinical Utility of a New Method to Identify Patients With Risk of Recurrent Colorectal Lesions and Personalization of Their Surveillance Based on Mutation Burden and Clinical-pathological Phenotype | 5 years
  To identify patients with high risk of metachronous colorectal lesions and try to design and optimal intervals of surveillance colonoscopies, especially in the high-risk group of patients, using mutation and clinical-pathologic phenotype.

SECONDARY OUTCOMES:
Determination of the mutation profile colorectal lesions | 5 years
  Determination of the mutation profile and mutation burden in 200 patients based on examination of all their index and synchronous lesions found during index colonoscopy using an established PCR/DCE-based heteroduplex method.
Mutational profil of colorectal lesions | 5 years
  Clinical and histopathological evaluation and mutational profiling of all metachronous lesions found during five-year surveillance period.

OTHER OUTCOMES:
Mutational phenotype of patient. | 5 years
  Correlation of clinical and histopathological parameters with mutational phenotype of patient.
Metachronous lesions | 5 years
  Correlation of patient's mutational phenotype with an occurrence of metachronous lesion/s during surveillance period.
Similarity of the mutation profile of lesions found in the same area | 5 years
  Analysis of the similarity of the mutation profile of lesions found in the same / close areas of the colorectum.

CONTACTS AND LOCATIONS:
Overall Officials: Stepan Suchanek, assoc. prof., Principal Investigator — Military University Hospital, Prague; Ondrej Ngo, Mgr., Study Director — Institute of Biostatistics and Analyses Brno; Lucie Benesova, RNDr., Study Director — Genomac Research Institute Prague; Ondrej Majek, RNDr., Study Chair — Institute of Biostatistics and Analyses Brno; Tereza Halkova, Mgr., Study Chair — Genomac Research Institute Prague
Locations (1):
- Military University Hospital, Prague, Czechia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Grega T, Kmochova K, Hejcmanova K, Ngo O, Brodyuk N, Majek O, Bures J, Urbanek P, Zavoral M, Suchanek S. Impact of narrow band imaging in prediction of histology of advanced colorectal neoplasia. Sci Rep. 2025 Jan 9;15(1):1414. doi: 10.1038/s41598-025-85669-w. PMID 39789214